CLINICAL TRIAL: NCT02897310
Title: Outcomes of Critically Ill Patients With Severe Acute Kidney Injury Requiring Renal Replacement Therapy
Acronym: PROVEER
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: PROVEER
Record Dates: First submitted 2016-08-19; First posted 2016-09-13 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Critical Illness; Acute Kidney Injury
Keywords: critically ill patients; acute kidney injury; renal replacement therapy; long term outcome
MeSH Terms: conditions — Critical Illness; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- critically ill patients: critically ill patients with acute kidney failure requiring renal replacement therapy

SUMMARY:
This study assess the vital status, renal function and renal recovery of patients admitted to intensive care unit and requiring renal replacement therapy for acute kidney failure. Patient follow up is up to 3 years after ICU admission when possible.

DETAILED DESCRIPTION:
Up to 50% of critically ill patients develop acute kidney injury and up to 10% require renal replacement therapy in the intensive care unit. This study aims to identify factors associated with mortality and to evaluate renal recovery of patients who had acute kidney failure requiring renal replacement therapy in intensive care unit at 1 and 3 years post intensive care unit admission.

ELIGIBILITY:
Inclusion Criteria:

* Adults admitted to the intensive care
* Acute kidney failure requiring renal replacement therapy

Exclusion Criteria:

* Patients suffering end stage renal failure requiring chronic renal replacement therapy
* Patients under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults hospitalised in intensive care and who developped acute renal failure requiring renal replacement therapy
Sampling Method: Probability Sample
Enrollment: 245 (Actual)
Dates: Start 2014-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
one-year mortality | year 1
  vital status

SECONDARY OUTCOMES:
hospital mortality | year 1
one year renal function | Year one

CONTACTS AND LOCATIONS:
Overall Officials: Aubron Cécile, Study Director — CHRU de Brest
Locations (1):
- CHRU de Brest, Brest, France